CLINICAL TRIAL: NCT06690047
Title: Treatment of Hereditary Angioedema Prodrome with Recombinant C1-esterase Inhibitor (Ruconest)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bernstein Clinical Research Center (Other)
Responsible Party: Principal Investigator, Jonathan A. Bernstein, MD, PI, Bernstein Clinical Research Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Ruc01
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Hereditary Angioedema
Keywords: prodrome
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — conestat alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ruconest (Active Comparator): open-label Ruconest
  Interventions: Biological: Ruconest
- No Ruconest (No Intervention): No Ruconest given

INTERVENTIONS:
Biological: Ruconest — recombinant human C1-esterase inhibitor
  Arms: Ruconest

SUMMARY:
To assess the efficacy of recombinant human C1-esterase inhibitor in the management of HAE prodrome for preventing the progression from prodrome to an acute angioedema attacks. Subjects will either receive Ruconest after the first 2 prodromes or during the last 2 prodromes. 5 clinic visits will occur within 24 hours of a prodrome. Subjects will complete prodrome severity and angioedema attack diaries

DETAILED DESCRIPTION:
After screening, subjects will be followed in the study for four consecutive prodromes. For prodromes designed to be treated with Ruconest, the drug will be administered within 12 hours of prodromal onset and prior to the onset of objective selling. Ruconset will be self-administered at home or by a healthcare professional at the recommended dose of 50 IU/kg body weight with maximum dose of 4200 IU as a slow IV injection over 5 minutes Subjects will be randomized into two arms after enrollment. Subjects in Arm A receives Ruconest after 1st and 2nd prodrome and no Ruconest after 3rd and 4th prodromes. Subjects in Arm B receive no Ruconest after 1st and 2nd prodrome and Ruconest after 3rd and 4th prodromes.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of HAE Type 1 and 2,
* One or more HAE attacks per month,
* History of 4 prodromes that proceed to angioedema attacks

Exclusion Criteria:

* History of thrombosis or arterial/venous thromboembolic attacks
* History of atherosclerosis, morbid obesity, immobility
* History of allergy to rabbits or products from rabbits
* History of life-threatening immediate allergic reactions to C1 esterase inhibitor preparations

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
The primary endpoint was the difference in response rates in preventing HAE attacks between Conestat Alfa®-treated vs. untreated HAE prodrome events. | up to 12 months from start of study
  A mixed model for repeated measures was used to determine the statistical significance of Conestat Alfa®'s clinical efficacy for treating the HAE prodrome versus the acute attack.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bernstein, MD, Principal Investigator — Bernstein Clinical Research Center
Locations (2):
- United States (2):
  - Clinical Research Center of Alabama, Birmingham, Alabama
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
not needed for manuscript